CLINICAL TRIAL: NCT04508088
Title: Skeletal Health and Bone Marrow Composition in Newly Diagnosed Adolescents With Crohn Disease
Status: Recruiting | Type: Observational
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Rebecca Gordon, MD, Rebecca Gordon, MD Attending Physician, Division of Pediatric Endocrinology, MGH; Assistant Professor of Pediatrics, Harvard Medical School, Massachusetts General Hospital
Other Study IDs: IRB-P00034878
Record Dates: First submitted 2020-07-22; First posted 2020-08-11 (Actual); Last update posted 2025-10-30 (Actual); Status verified 2025-10

CONDITIONS: Inflammatory Bowel Disease; Crohn Disease
Keywords: Crohn; Bone Marrow; Dual-energy X-ray absorptiometry; Peripheral Quantitative Computed Tomography; Magnetic Resonance Imaging
MeSH Terms: conditions — Inflammatory Bowel Diseases; Crohn Disease | interventions — Positron-Emission Tomography; Blood Specimen Collection

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — A) Bone turnover markers: We will assess markers of bone formation, including osteocalcin (OC) and procollagen type 1 N-terminal propeptide (P1NP), and a marker of bone resorption, c-telopeptide (CTX).
  B) Immune studies: We will first employ bulk RNA-seq on peripheral blood to evaluate molecular gene signatures that correlate with the various bone imaging phenotypes. Molecular markers that correlate with the bone imaging phenotypes will be used to inform development and validation of a CyTOF panel that will be used on matched PBMC samples. Utilizing CyTOF, we will evaluate differences in immune cellular populations between CD patients with normal versus low BMD, and matched controls.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Crohn Disease: This group will be 46 adolescents, ages 13-20, who have been recently (within 3 months) diagnosed with Crohn Disease.
  All participants will have a two study visits approximately one year apart during which the listed diagnostic testing will be performed.
  Interventions: Diagnostic Test: Coronal T1 weighted spin echo images; Diagnostic Test: Spin-lattice relaxation (T1); Diagnostic Test: Magnetic resonance spectroscopy; Diagnostic Test: Blood Draw
- Control: Controls will be matched for age, Tanner staging, and BMI percentile.
  All participants will have a two study visits approximately one year apart during which the listed diagnostic testing will be performed.
  Interventions: Diagnostic Test: Coronal T1 weighted spin echo images; Diagnostic Test: Spin-lattice relaxation (T1); Diagnostic Test: Magnetic resonance spectroscopy; Diagnostic Test: Blood Draw

INTERVENTIONS:
Diagnostic Test: Coronal T1 weighted spin echo images — Coronal T1 weighted spin echo images will be obtained through the knee with a field of view of 16cm to include distal femoral and proximal tibial metaphyses.
Diagnostic Test: Spin-lattice relaxation (T1) — Spin-lattice relaxation (T1) relaxometry acquisition consisting of seven fast spin echo (FSE) acquisitions through the knee. T1 maps from the T1 relaxometry images will be generated using a two-parameter-fit iterative algorithm developed in-house using IDL software (Harris Geospatial Solutions, Melbourne, FL, USA). Mean T1 values for each region will be recorded. The anatomical locations of these regions will be consistent in size for all subjects and location. The locations chosen for the primary endpoints are ones that are known to be rich in red and yellow marrow, respectively.
Diagnostic Test: Magnetic resonance spectroscopy — Magnetic resonance spectroscopy. MRS will be performed within a 1 mL voxel situated in the medial aspect of the distal femoral metaphysis. A single voxel point resolved spectral acquisition (PRESS) technique will be used to acquire non-water suppressed spectra at echo times of 20, 30, 40, and 50 ms using 32 signal averages per echo time with a TR of 2.5 s (total scan time = 5.4 minutes). Spectral fits using JMRUI MRS processing software (www.jmrui.eu) to the water and methylene/methyl resonances will be used to quantify peak areas and establish T2 corrected fat/(fat + water) ratios.
Diagnostic Test: Blood Draw — Blood draw. Blood draws will be used to attain and assess markers of bone formation/resorption and to perform immune studies. Specific markers of bone formation that will be assessed include osteocalcin (OC) and procollagen type 1 N-terminal propeptide (P1NP), and a marker of bone resorption, c-telopeptide (CTX). We will also evaluate molecular gene signatures from the blood samples that correlate with the previously described bone imaging phenotypes. At that point, the information will be used to develop a CyTOF panel to evaluate differences in immune cellular populations between CD patients with normal versus low BMD, and matched controls.

SUMMARY:
The investigators will be evaluating bone marrow composition via magnetic resonance imaging in newly diagnosed adolescents with Crohn disease (CD) compared to healthy, matched controls. The investigators will also be assessing their bone mineral density via other imaging modalities, including dual-energy X-ray absorptiometry and peripheral quantitative computed tomography. This longitudinal project will focus on abnormalities in bone marrow composition, and specifically whether adolescents with newly diagnosed CD exhibit increased bone marrow fat, its association with bone mineral density (BMD) and the underlying pathophysiology, including bone turnover markers and immune cellular/molecular parameters.

DETAILED DESCRIPTION:
Less than optimal bone health has been seen in children that have inflammatory bowel disease (IBD), including Crohn disease (CD). This can present as low bone density or altered bone structure, weakening the bones and increasing fragility and fracture risk. As adolescence is especially important in bone development, conditions such as CD during this time can lead to long term bone issues. The underlying mechanisms are not well understood, but what is known is that red bone marrow converts to fat-rich yellow marrow. This study aims to focus on abnormalities in bone marrow, and specifically whether adolescents who have been diagnosed with CD have more bone marrow fat.

The primary hypothesis is that newly diagnosed CD is associated with increased fat levels in bone, which is associated with decreased bone formation and suboptimal bone health. The central objective is to obtain longitudinal data on the differences in bone marrow between healthy adolescents and those with CD. Long term, the investigators want to study how abnormal fat tissue and suboptimal bone health relate to each other.

The study involves 46 adolescents recently diagnosed with CD and 46 healthy adolescents. Eligibility criteria include no other chronic diseases that affect bone health and limited use of bone altering medications in the last three months. The CD adolescents will be matched with healthy adolescents based on age, stage of puberty, and BMI percentile. Additional data on CD participants will be collected via a chart review that will enable us to more fully characterize their CD.

Imaging will include MRIs of the knee. Measurements will include a visual assessment and quantitative marrow fat analysis, dual-energy X-ray absorptiometry (DXA), and peripheral quantitative computed tomography (pQCT). All scans will be for research purposes only. The MRIs will be evaluated for any abnormalities, and if there is an incidental finding, it will be reported to the primary care physician.

Additionally, blood draws will be used to attain and assess markers of bone formation/resorption and to perform immune studies.

ELIGIBILITY:
Inclusion Criteria:

* Crohn's Disease diagnosed within the past 3 months, or a healthy, matched control

Exclusion Criteria:

* Participants with chronic disease known to affect skeletal metabolism
* Participants on certain medications within the prior 3 months that are known to affect skeletal metabolism
* Participants who are pregnant
* Participants who have a history of: claustrophobia, internal body metal that is not compatible with MRI machine, or a known abnormality on or adjacent to the left knee

Ages: 13 Years to 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: The experimental group will be adolescents aged 13-20 with newly diagnosed CD (within 3 months of diagnosis, based on histologic diagnosis and verified with their gastroenterologist).
  The control group will be matched for age (within 1 year), pubertal stage (based on Tanner staging), and BMI percentile. Tanner staging will be based on clinically documented Tanner stage by GI physician for participants with CD and by their primary care physician for control participants. If there is no documented Tanner staging, then it will either be performed by the participants primary care physician, or by a pediatric endocrinologist.
Sampling Method: Non-Probability Sample
Enrollment: 92 (Estimated)
Dates: Start 2020-09-10 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Bone marrow adiposity by magnetic resonance imaging (MRI) | Baseline and One Year follow-up
  Change in Bone marrow adiposity measured by MRI (T1 maps)
Magnetic resonance spectroscopy (MRS) | Baseline and One Year follow-up
  Change in T2 corrected fat/(fat+ water) ratios

SECONDARY OUTCOMES:
Total body bone mineral density Z-score by Dual-energy X-ray absorptiometry (DXA) | Baseline and One Year follow-up
  Change in Total body BMD Z-score
Spine BMD Z-score by DXA | Baseline and One Year follow-up
  Change in Lumbar spine BMD Z-score
Spine apparent density Z-score by DXA | Baseline and One Year follow-up
  Change in Lumbar spine bone mineral apparent density (g/cm3)
Volumetric bone mineral density (vBMD) | Baseline and One Year follow-up
  Change in Quantitative computed tomography (pQCT) scans will be obtained at sites 3%, 38%, and 66% of tibial length proximal to the distal growth plate
Bone strength by quantitative computed tomography pQCT | Baseline and One Year follow-up
  Change in PQCT scans will be obtained at sites 3%, 38%, and 66% of tibial length proximal to the distal growth plate
Bone Formation Marker #1 | Baseline and One Year follow-up
  Change in bone formation assessed by osteocalcin (ng/mL)
Bone Formation Marker #2 | Baseline and One Year follow-up
  Change in bone formation assessed by procollagen type 1 N-terminal propeptide (ng/mL)
Bone Resorption Marker | Baseline and One Year follow-up
  Change in bone resorption assessed by c-telopeptide (pg/ml)
Immune Studies | Baseline and One Year follow-up
  Bulk RNA-sequencing on peripheral blood to evaluate molecular gene signatures that correlate with various bone imaging phenotypes; these will then be used to inform development and validation of a Mass Cytometry by Time-of-Flight panel that will be used on matched peripheral blood mononuclear cells samples.
Current Crohn's Disease Activity | Baseline and One Year follow-up
  Current Crohn's disease activity will be assessed using the pediatric Crohn disease activity index (PCDAI). The assessment will be made based on questionnaires answered.
Physical Activity | Baseline and One Year follow-up
  Physical activity will be assessed through a physical activity questionnaire
Dietary Calcium Intake | Baseline and One Year follow-up
  Dietary calcium intake will be assessed through a targeted dietary questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca Gordon, MD, Principal Investigator — Boston Children's Hospital
Locations (1):
- Boston Children's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gupta A, Paski S, Issenman R, Webber C. Lumbar spine bone mineral density at diagnosis and during follow-up in children with IBD. J Clin Densitom. 2004 Fall;7(3):290-5. doi: 10.1385/jcd:7:3:290. PMID 15319499
- [Background] Sylvester FA, Wyzga N, Hyams JS, Davis PM, Lerer T, Vance K, Hawker G, Griffiths AM. Natural history of bone metabolism and bone mineral density in children with inflammatory bowel disease. Inflamm Bowel Dis. 2007 Jan;13(1):42-50. doi: 10.1002/ibd.20006. PMID 17206638
- [Background] Schmidt S, Mellstrom D, Norjavaara E, Sundh SV, Saalman R. Low bone mineral density in children and adolescents with inflammatory bowel disease: a population-based study from Western Sweden. Inflamm Bowel Dis. 2009 Dec;15(12):1844-50. doi: 10.1002/ibd.20962. Epub 2009 Apr 30. PMID 19408319
- [Background] Werkstetter KJ, Pozza SB, Filipiak-Pittroff B, Schatz SB, Prell C, Bufler P, Koletzko B, Koletzko S. Long-term development of bone geometry and muscle in pediatric inflammatory bowel disease. Am J Gastroenterol. 2011 May;106(5):988-98. doi: 10.1038/ajg.2010.495. Epub 2011 Jan 11. PMID 21224841
- [Background] Bechtold S, Alberer M, Arenz T, Putzker S, Filipiak-Pittroff B, Schwarz HP, Koletzko S. Reduced muscle mass and bone size in pediatric patients with inflammatory bowel disease. Inflamm Bowel Dis. 2010 Feb;16(2):216-25. doi: 10.1002/ibd.21021. PMID 19637389
- [Background] Dubner SE, Shults J, Baldassano RN, Zemel BS, Thayu M, Burnham JM, Herskovitz RM, Howard KM, Leonard MB. Longitudinal assessment of bone density and structure in an incident cohort of children with Crohn's disease. Gastroenterology. 2009 Jan;136(1):123-30. doi: 10.1053/j.gastro.2008.09.072. Epub 2008 Nov 1. PMID 19026647
- [Background] Bonjour JP, Theintz G, Law F, Slosman D, Rizzoli R. Peak bone mass. Osteoporos Int. 1994;4 Suppl 1:7-13. doi: 10.1007/BF01623429. PMID 8081064
- [Background] Tuchman S, Thayu M, Shults J, Zemel BS, Burnham JM, Leonard MB. Interpretation of biomarkers of bone metabolism in children: impact of growth velocity and body size in healthy children and chronic disease. J Pediatr. 2008 Oct;153(4):484-90. doi: 10.1016/j.jpeds.2008.04.028. Epub 2008 Jun 16. PMID 18555484
- [Background] Waitches G, Zawin JK, Poznanski AK. Sequence and rate of bone marrow conversion in the femora of children as seen on MR imaging: are accepted standards accurate? AJR Am J Roentgenol. 1994 Jun;162(6):1399-406. doi: 10.2214/ajr.162.6.8192007.
- [Background] Taccone A, Oddone M, Dell'Acqua AD, Occhi M, Ciccone MA. MRI "road-map" of normal age-related bone marrow. II. Thorax, pelvis and extremities. Pediatr Radiol. 1995;25(8):596-606. doi: 10.1007/BF02011826. PMID 8570312
- [Background] Taccone A, Oddone M, Occhi M, Dell'Acqua AD, Ciccone MA. MRI "road-map" of normal age-related bone marrow. I. Cranial bone and spine. Pediatr Radiol. 1995;25(8):588-95. doi: 10.1007/BF02011825. PMID 8570311
- [Background] Thayu M, Leonard MB, Hyams JS, Crandall WV, Kugathasan S, Otley AR, Olson A, Johanns J, Marano CW, Heuschkel RB, Veereman-Wauters G, Griffiths AM, Baldassano RN; Reach Study Group. Improvement in biomarkers of bone formation during infliximab therapy in pediatric Crohn's disease: results of the REACH study. Clin Gastroenterol Hepatol. 2008 Dec;6(12):1378-84. doi: 10.1016/j.cgh.2008.07.010. PMID 19081527
- [Background] Thornton D, Gordon CM. Restrictive Eating Disorders and Skeletal Health in Adolescent Girls and Young Women. Calcif Tissue Int. 2017 May;100(5):449-460. doi: 10.1007/s00223-016-0164-0. Epub 2016 Jun 23. PMID 27339670
- [Background] Ecklund K, Vajapeyam S, Feldman HA, Buzney CD, Mulkern RV, Kleinman PK, Rosen CJ, Gordon CM. Bone marrow changes in adolescent girls with anorexia nervosa. J Bone Miner Res. 2010 Feb;25(2):298-304. doi: 10.1359/jbmr.090805. PMID 19653811
- [Background] Ecklund K, Vajapeyam S, Mulkern RV, Feldman HA, O'Donnell JM, DiVasta AD, Gordon CM. Bone marrow fat content in 70 adolescent girls with anorexia nervosa: Magnetic resonance imaging and magnetic resonance spectroscopy assessment. Pediatr Radiol. 2017 Jul;47(8):952-962. doi: 10.1007/s00247-017-3856-3. Epub 2017 Apr 22. PMID 28432403
- [Background] Meunier P, Aaron J, Edouard C, Vignon G. Osteoporosis and the replacement of cell populations of the marrow by adipose tissue. A quantitative study of 84 iliac bone biopsies. Clin Orthop Relat Res. 1971 Oct;80:147-54. doi: 10.1097/00003086-197110000-00021. No abstract available. PMID 5133320
- [Background] Yeung DK, Griffith JF, Antonio GE, Lee FK, Woo J, Leung PC. Osteoporosis is associated with increased marrow fat content and decreased marrow fat unsaturation: a proton MR spectroscopy study. J Magn Reson Imaging. 2005 Aug;22(2):279-85. doi: 10.1002/jmri.20367. PMID 16028245
- [Background] Griffith JF, Yeung DK, Antonio GE, Lee FK, Hong AW, Wong SY, Lau EM, Leung PC. Vertebral bone mineral density, marrow perfusion, and fat content in healthy men and men with osteoporosis: dynamic contrast-enhanced MR imaging and MR spectroscopy. Radiology. 2005 Sep;236(3):945-51. doi: 10.1148/radiol.2363041425. Epub 2005 Jul 29. PMID 16055699
- [Background] Shen W, Chen J, Punyanitya M, Shapses S, Heshka S, Heymsfield SB. MRI-measured bone marrow adipose tissue is inversely related to DXA-measured bone mineral in Caucasian women. Osteoporos Int. 2007 May;18(5):641-7. doi: 10.1007/s00198-006-0285-9. Epub 2006 Dec 1. PMID 17139464
- [Background] Bredella MA, Fazeli PK, Miller KK, Misra M, Torriani M, Thomas BJ, Ghomi RH, Rosen CJ, Klibanski A. Increased bone marrow fat in anorexia nervosa. J Clin Endocrinol Metab. 2009 Jun;94(6):2129-36. doi: 10.1210/jc.2008-2532. Epub 2009 Mar 24. PMID 19318450
- [Background] Botolin S, McCabe LR. Bone loss and increased bone adiposity in spontaneous and pharmacologically induced diabetic mice. Endocrinology. 2007 Jan;148(1):198-205. doi: 10.1210/en.2006-1006. Epub 2006 Oct 19. PMID 17053023
- [Background] Saha MT, Sievanen H, Salo MK, Tulokas S, Saha HH. Bone mass and structure in adolescents with type 1 diabetes compared to healthy peers. Osteoporos Int. 2009 Aug;20(8):1401-6. doi: 10.1007/s00198-008-0810-0. Epub 2008 Dec 13. PMID 19083073
- [Background] Maggio AB, Ferrari S, Kraenzlin M, Marchand LM, Schwitzgebel V, Beghetti M, Rizzoli R, Farpour-Lambert NJ. Decreased bone turnover in children and adolescents with well controlled type 1 diabetes. J Pediatr Endocrinol Metab. 2010 Jul;23(7):697-707. doi: 10.1515/jpem.2010.23.7.697. PMID 20857842
- [Background] Gunczler P, Lanes R, Paoli M, Martinis R, Villaroel O, Weisinger JR. Decreased bone mineral density and bone formation markers shortly after diagnosis of clinical type 1 diabetes mellitus. J Pediatr Endocrinol Metab. 2001 May;14(5):525-8. doi: 10.1515/jpem.2001.14.5.525. PMID 11393573
- [Background] Vives-Pi M, Somoza N, Fernandez-Alvarez J, Vargas F, Caro P, Alba A, Gomis R, Labeta MO, Pujol-Borrell R. Evidence of expression of endotoxin receptors CD14, toll-like receptors TLR4 and TLR2 and associated molecule MD-2 and of sensitivity to endotoxin (LPS) in islet beta cells. Clin Exp Immunol. 2003 Aug;133(2):208-18. doi: 10.1046/j.1365-2249.2003.02211.x. PMID 12869026
- [Background] Liu D, Cardozo AK, Darville MI, Eizirik DL. Double-stranded RNA cooperates with interferon-gamma and IL-1 beta to induce both chemokine expression and nuclear factor-kappa B-dependent apoptosis in pancreatic beta-cells: potential mechanisms for viral-induced insulitis and beta-cell death in type 1 diabetes mellitus. Endocrinology. 2002 Apr;143(4):1225-34. doi: 10.1210/endo.143.4.8737. PMID 11897677
- [Background] Willcox A, Richardson SJ, Bone AJ, Foulis AK, Morgan NG. Analysis of islet inflammation in human type 1 diabetes. Clin Exp Immunol. 2009 Feb;155(2):173-81. doi: 10.1111/j.1365-2249.2008.03860.x. PMID 19128359
- [Background] Braidotti P, Stagni L. A critical damping approach for assessing the role of marrow fat on the mechanical strength of trabecular bone. Med Hypotheses. 2007;69(1):43-6. doi: 10.1016/j.mehy.2006.09.074. Epub 2007 Feb 6. PMID 17287095
- [Background] Schellinger D, Lin CS, Lim J, Hatipoglu HG, Pezzullo JC, Singer AJ. Bone marrow fat and bone mineral density on proton MR spectroscopy and dual-energy X-ray absorptiometry: their ratio as a new indicator of bone weakening. AJR Am J Roentgenol. 2004 Dec;183(6):1761-5. doi: 10.2214/ajr.183.6.01831761. PMID 15547224
- [Background] Pittenger MF, Mackay AM, Beck SC, Jaiswal RK, Douglas R, Mosca JD, Moorman MA, Simonetti DW, Craig S, Marshak DR. Multilineage potential of adult human mesenchymal stem cells. Science. 1999 Apr 2;284(5411):143-7. doi: 10.1126/science.284.5411.143. PMID 10102814
- [Background] Tontonoz P, Hu E, Graves RA, Budavari AI, Spiegelman BM. mPPAR gamma 2: tissue-specific regulator of an adipocyte enhancer. Genes Dev. 1994 May 15;8(10):1224-34. doi: 10.1101/gad.8.10.1224. PMID 7926726
- [Background] Tontonoz P, Hu E, Spiegelman BM. Stimulation of adipogenesis in fibroblasts by PPAR gamma 2, a lipid-activated transcription factor. Cell. 1994 Dec 30;79(7):1147-56. doi: 10.1016/0092-8674(94)90006-x. PMID 8001151
- [Background] Hassan MQ, Tare RS, Lee SH, Mandeville M, Morasso MI, Javed A, van Wijnen AJ, Stein JL, Stein GS, Lian JB. BMP2 commitment to the osteogenic lineage involves activation of Runx2 by DLX3 and a homeodomain transcriptional network. J Biol Chem. 2006 Dec 29;281(52):40515-26. doi: 10.1074/jbc.M604508200. Epub 2006 Oct 23. PMID 17060321
- [Background] Gaur T, Lengner CJ, Hovhannisyan H, Bhat RA, Bodine PV, Komm BS, Javed A, van Wijnen AJ, Stein JL, Stein GS, Lian JB. Canonical WNT signaling promotes osteogenesis by directly stimulating Runx2 gene expression. J Biol Chem. 2005 Sep 30;280(39):33132-40. doi: 10.1074/jbc.M500608200. Epub 2005 Jul 25. PMID 16043491
- [Background] Beresford JN, Bennett JH, Devlin C, Leboy PS, Owen ME. Evidence for an inverse relationship between the differentiation of adipocytic and osteogenic cells in rat marrow stromal cell cultures. J Cell Sci. 1992 Jun;102 ( Pt 2):341-51. doi: 10.1242/jcs.102.2.341. PMID 1400636
- [Background] Lecka-Czernik B, Moerman EJ, Grant DF, Lehmann JM, Manolagas SC, Jilka RL. Divergent effects of selective peroxisome proliferator-activated receptor-gamma 2 ligands on adipocyte versus osteoblast differentiation. Endocrinology. 2002 Jun;143(6):2376-84. doi: 10.1210/endo.143.6.8834. PMID 12021203
- [Background] Gimble JM, Morgan C, Kelly K, Wu X, Dandapani V, Wang CS, Rosen V. Bone morphogenetic proteins inhibit adipocyte differentiation by bone marrow stromal cells. J Cell Biochem. 1995 Jul;58(3):393-402. doi: 10.1002/jcb.240580312. PMID 7593260
- [Background] Akune T, Ohba S, Kamekura S, Yamaguchi M, Chung UI, Kubota N, Terauchi Y, Harada Y, Azuma Y, Nakamura K, Kadowaki T, Kawaguchi H. PPARgamma insufficiency enhances osteogenesis through osteoblast formation from bone marrow progenitors. J Clin Invest. 2004 Mar;113(6):846-55. doi: 10.1172/JCI19900. PMID 15067317
- [Background] Vajapeyam S, Ecklund K, Mulkern RV, Feldman HA, O'Donnell JM, DiVasta AD, Rosen CJ, Gordon CM. Magnetic resonance imaging and spectroscopy evidence of efficacy for adrenal and gonadal hormone replacement therapy in anorexia nervosa. Bone. 2018 May;110:335-342. doi: 10.1016/j.bone.2018.02.021. Epub 2018 Feb 26. PMID 29496516
- [Background] Moore SG, Dawson KL. Red and yellow marrow in the femur: age-related changes in appearance at MR imaging. Radiology. 1990 Apr;175(1):219-23. doi: 10.1148/radiology.175.1.2315484.
- [Background] Ricci C, Cova M, Kang YS, Yang A, Rahmouni A, Scott WW Jr, Zerhouni EA. Normal age-related patterns of cellular and fatty bone marrow distribution in the axial skeleton: MR imaging study. Radiology. 1990 Oct;177(1):83-8. doi: 10.1148/radiology.177.1.2399343.
- [Background] Carter DR, Bouxsein ML, Marcus R. New approaches for interpreting projected bone densitometry data. J Bone Miner Res. 1992 Feb;7(2):137-45. doi: 10.1002/jbmr.5650070204. PMID 1570758
- [Background] Kalkwarf HJ, Zemel BS, Gilsanz V, Lappe JM, Horlick M, Oberfield S, Mahboubi S, Fan B, Frederick MM, Winer K, Shepherd JA. The bone mineral density in childhood study: bone mineral content and density according to age, sex, and race. J Clin Endocrinol Metab. 2007 Jun;92(6):2087-99. doi: 10.1210/jc.2006-2553. Epub 2007 Feb 20. PMID 17311856
- [Background] Shepherd JA, Wang L, Fan B, Gilsanz V, Kalkwarf HJ, Lappe J, Lu Y, Hangartner T, Zemel BS, Fredrick M, Oberfield S, Winer KK. Optimal monitoring time interval between DXA measures in children. J Bone Miner Res. 2011 Nov;26(11):2745-52. doi: 10.1002/jbmr.473. PMID 21773995
- [Background] Leonard MB, Elmi A, Mostoufi-Moab S, Shults J, Burnham JM, Thayu M, Kibe L, Wetzsteon RJ, Zemel BS. Effects of sex, race, and puberty on cortical bone and the functional muscle bone unit in children, adolescents, and young adults. J Clin Endocrinol Metab. 2010 Apr;95(4):1681-9. doi: 10.1210/jc.2009-1913. Epub 2010 Feb 15. PMID 20157194
- [Background] Thayu M, Shults J, Burnham JM, Zemel BS, Baldassano RN, Leonard MB. Gender differences in body composition deficits at diagnosis in children and adolescents with Crohn's disease. Inflamm Bowel Dis. 2007 Sep;13(9):1121-8. doi: 10.1002/ibd.20149. PMID 17427245
- [Background] Augat P, Reeb H, Claes LE. Prediction of fracture load at different skeletal sites by geometric properties of the cortical shell. J Bone Miner Res. 1996 Sep;11(9):1356-63. doi: 10.1002/jbmr.5650110921. PMID 8864911
- [Background] Liu D, Manske SL, Kontulainen SA, Tang C, Guy P, Oxland TR, McKay HA. Tibial geometry is associated with failure load ex vivo: a MRI, pQCT and DXA study. Osteoporos Int. 2007 Jul;18(7):991-7. doi: 10.1007/s00198-007-0325-0. Epub 2007 Feb 1. PMID 17268944
- [Background] Kanal E, Barkovich AJ, Bell C, Borgstede JP, Bradley WG Jr, Froelich JW, Gilk T, Gimbel JR, Gosbee J, Kuhni-Kaminski E, Lester JW Jr, Nyenhuis J, Parag Y, Schaefer DJ, Sebek-Scoumis EA, Weinreb J, Zaremba LA, Wilcox P, Lucey L, Sass N; ACR Blue Ribbon Panel on MR Safety. ACR guidance document for safe MR practices: 2007. AJR Am J Roentgenol. 2007 Jun;188(6):1447-74. doi: 10.2214/AJR.06.1616. No abstract available. PMID 17515363
- [Background] Thomas SR, Kalkwarf HJ, Buckley DD, Heubi JE. Effective dose of dual-energy X-ray absorptiometry scans in children as a function of age. J Clin Densitom. 2005 Winter;8(4):415-22. doi: 10.1385/jcd:8:4:415. PMID 16311426
- [Background] Harris PA, Taylor R, Thielke R, Payne J, Gonzalez N, Conde JG. Research electronic data capture (REDCap)--a metadata-driven methodology and workflow process for providing translational research informatics support. J Biomed Inform. 2009 Apr;42(2):377-81. doi: 10.1016/j.jbi.2008.08.010. Epub 2008 Sep 30. PMID 18929686
- [Background] Mitsialis V, Wall S, Liu P, Ordovas-Montanes J, Parmet T, Vukovic M, Spencer D, Field M, McCourt C, Toothaker J, Bousvaros A; Boston Children's Hospital Inflammatory Bowel Disease Center; Brigham and Women's Hospital Crohn's and Colitis Center; Shalek AK, Kean L, Horwitz B, Goldsmith J, Tseng G, Snapper SB, Konnikova L. Single-Cell Analyses of Colon and Blood Reveal Distinct Immune Cell Signatures of Ulcerative Colitis and Crohn's Disease. Gastroenterology. 2020 Aug;159(2):591-608.e10. doi: 10.1053/j.gastro.2020.04.074. Epub 2020 May 16. PMID 32428507
- [Background] Sigurdsson GV, Schmidt S, Mellstrom D, Ohlsson C, Kindblom JM, Lorentzon M, Saalman R. Bone Mass Development from Childhood into Young Adulthood in Patients with Childhood-onset Inflammatory Bowel Disease. Inflamm Bowel Dis. 2017 Dec;23(12):2215-2226. doi: 10.1097/MIB.0000000000001277. PMID 29064856